CLINICAL TRIAL: NCT02342119
Title: Increasing Equity in Transplant Evaluation and Living Donor Kidney Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Mary Amanda Dew, Mary Amanda Dew, PhD, Professor of Psychiatry, Psychology, Epidemiology, Biostatistics, and Clinical and Translational Science, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PRO13100511; 5R01DK101715-04 (NIH)
Record Dates: First submitted 2015-01-07; First posted 2015-01-19 (Estimated); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: End-stage Kidney Disease
Keywords: kidney transplantation; race disparities; living donor kidney transplantation; transplant evaluation
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- KTFT+TALK (Experimental): Patients who are being evaluated for a kidney transplantation via Kidney Transplant Fast Track and who are receiving the Talking About Living Kidney Donation intervention
  Interventions: Other: Talking About Living Kidney Donation; Other: Kidney Transplant Fast Track
- KTFT+No TALK (Active Comparator): Patients who are being evaluated for a kidney transplantation via Kidney Transplant Fast Track and who are not receiving the Talking About Living Kidney Donation intervention
  Interventions: Other: Kidney Transplant Fast Track

INTERVENTIONS:
Other: Talking About Living Kidney Donation — TALK participants receive a culturally sensitive educational booklet and video. A study interventionist encourages participants to share the materials with their family members or friends. Materials provide information to encourage patient and families shared and informed consideration of LDKT, including: 1) information about eligibility for LDKT, 2) the clinical evaluation required for LDKT, 3) the donor selection process, 4) surgical procedures for transplantation and donation, 5), and concerns brought forth about these factors, identified through structured group interviews.
  Other Names: TALK
  Arms: KTFT+TALK
Other: Kidney Transplant Fast Track — KTFT is a one-day streamlined transplant evaluation process. Every patient who is evaluated at the University of Pittsburgh Starzl Transplant Center receives the KTFT. This approach involves completion of most or all testing on the same day that patients arrive for their first pre-transplant clinic appointment, rather than providing them with a list of tests they complete on their own with their referring physician. If patients are unable to be scheduled the same day, the transplant clinic scheduler secures appointment times and preparatory material for all testing to be completed within a 2 week period.
  Other Names: KTFT

SUMMARY:
Living donor kidney transplantation (LDKT) is the optimal treatment for end-stage kidney disease (ESKD). But, the evaluation process for a kidney transplant is lengthy, time consuming, and burdensome to the patient. Also, race disparities exist in rates of transplant evaluation completion, transplantation, and LDKT. Our previous and ongoing NIDDK-funded research indicates that cultural factors (i.e., perceived discrimination in health care, religious objection to LDKT), transplant knowledge, and demographic characteristics (e.g., age, education, income) independently and significantly predict time to complete transplant evaluation. In December 2012 the investigators' transplant center implemented a one-day streamlined evaluation process, dubbed Kidney Transplant Fast Track (KTFT), but it has not been evaluated for efficacy or cost effectiveness. Thus, the investigators propose a quasi-experiment to determine the efficacy and cost-effectiveness of the KTFT (n=1030) compared to historical controls (n=1140) who were recruited for the investigators' current NIDDK study to increase transplant rates. At the same time, the investigators will conduct a randomized controlled trial (RCT) targeting vulnerable patients with the educational component of the TALK intervention (Talking About Live Kidney Donation) to increase LDKT. For both components of the proposal, the investigators will target vulnerable populations because they are most at risk for extended evaluation times and lower rates of LDKT. Using CONSORT standards, participants will be randomly assigned to TALK (n=515) versus no-TALK (n=515) conditions and undergo two interviews at pre-transplant work-up and at completion of transplant evaluation in order to: (1) test whether KTFT and TALK will reduce transplant evaluation time, and increase rates of transplant and LDKT in members of vulnerable groups; (2) determine whether engaging in a streamlined and coordinated-care evaluation experience within the transplant center reduces negative perceptions of the healthcare system; and (3) test the cost effectiveness of the KTFT with TALK relative to standard practices. The results of this two-pronged approach will help pave the way for other transplant centers to implement a fast-track system at their sites, improve quality of care by transplanting a larger number of vulnerable patients, and may help address stark race/ethnic disparities in rates of LDKT.

DETAILED DESCRIPTION:
SPECIFIC AIMS Kidney transplantation (KT) is the optimal treatment for end-stage kidney disease (ESKD). It reduces mortality, improves quality of life, and is less costly than dialysis. Further, living donor KT (LDKT) is better than deceased donor KT (DDKT) because: (a) patients who can identify a living donor will get a KT much more quickly than ones awaiting DDKT and, (b) LDKT yields better outcomes than DDKT by improving cost effectiveness, reducing morbidity, and increasing long-term survival. The KT evaluation process, which occurs after patients have been referred for KT, is lengthy, time consuming, and burdensome to the patient. It requires patients to complete numerous tests (e.g., blood work, cardiac checks, pap smear, etc.) in order to be presented to the transplant team and accepted for KT. Although some variation between centers exists, typically patients must complete testing on their own, and ensure that their clinical providers forward results to the transplant team. This requires significant oversight and follow-up by the patient with each clinical provider.

The investigators' previous and ongoing NIDDK-funded research indicates that cultural factors (i.e., perceived discrimination in health care, religious objection to LDKT), KT knowledge, and demographic characteristics (e.g., age, education, income) independently and significantly predict time to complete KT evaluation. Similarly, the investigators' research found that African Americans (AA) take significantly longer to complete the evaluation process, and that the factors identified to predict longer time to complete evaluation are significantly associated with race. Other research has shown significant disparities in ESKD and its treatment for members of vulnerable groups (e.g., Hispanic/Latino, Native Americans, low income), and that African Americans (AA) are a particularly vulnerable group. For example, although ESKD in AA is four times greater than in whites (WH), AA are less than half as likely to undergo KT. AA race is associated with: (a) a longer time to complete evaluation for KT,19 (b) lower likelihood of getting a KT, (c) lower rates of pre-emptive listing for KT, and, (d) lower rates of LDKT versus DDKT. Therefore, two of the best ways to reduce disparities in KT may be to increase (a) the number of vulnerable group members who complete KT evaluation and (b) the rate of LDKT. This study is a two-pronged approach to address these two critical areas.

In December 2012 the investigators' transplant center implemented a one-day streamlined evaluation process, which they dubbed Kidney Transplant Fast Track (KTFT), but it has not been evaluated for efficacy or cost effectiveness. Thus, the investigators propose a quasi-experiment to determine the efficacy and cost-effectiveness in vulnerable groups of the KTFT compared to historical controls who were recruited for their previous NIDDK study. This component of the study will allow the investigators to take advantage of a unique and unusual natural experiment which occurred due to system-level clinical changes in the way patients are evaluated for KT at their center. The investigators will test if KTFT yields faster evaluation completion times, and ultimately higher KT rates. The second component of this study is to conduct a randomized controlled trial (RCT) targeting KTFT patients with the educational component of the TALK intervention to increase LDKT. The KT evaluation period poses an excellent opportunity to encourage patients to pursue LDKT. However, if the evaluation period is compressed via programs such as KTFT, it becomes critical to maximize patients' ability to pursue LDKT. For both the quasi-experimental and RCT components of this work, the investigators will target vulnerable populations because they are most at risk for extended evaluation times and lower rates of LDKT and these are the two most critical factors leading to disparities in KT. Specifically, the investigators intend to:

SA1: Test the efficacy and cost-effectiveness of a comprehensive, system-level fast-track KT evaluation for vulnerable groups in reducing time to complete KT evaluation, and increasing KT rates.

H1a: Compared to historical controls, evaluation time will be reduced with KTFT evaluation.

H1b: Compared to historical controls, KTFT will increase KT rates. H1c: KTFT will be a cost-effective evaluation strategy relative to standard evaluation practices.

SA2: Using an RCT, test the effectiveness of the TALK intervention in increasing rates of LDKT during KTFT.

H2a: Compared to the no-TALK controls, rates of LDKT will be higher in the TALK group.

H2b: Participants in KTFT+TALK will have higher KT rates than historical controls and no-TALK controls.

H2c: The addition of KTFT+TALK will be a cost-effective strategy to increase LDKT rates.

SA3: Determine whether engaging in a comprehensive, streamlined, and coordinated-care evaluation experience within the transplant center reduces negative perceptions of the healthcare system.

H3a: After KTFT, participants will report lower levels of medical mistrust than before KTFT, and lower than historical controls.

H3b: After KTFT, AA participants will report lower levels of perceived discrimination and racism than before KTFT, and lower than historical controls.

RESEARCH STRATEGY

SIGNIFICANCE The incidence and prevalence of end-stage kidney disease (ESKD) cases in the US nearly doubled in the 1990s. In the US population, more than 590,000 adults are currently treated for ESKD, and another 7.4 million have chronic kidney disease, which typically advances to ESKD. The aging of baby boomers, changing racial distributions, and increasing prevalence of diabetes in the US indicates that the prevalence of ESKD will continue to rise. In 2010, the US spent more than $27 billion in Medicare funds to treat patients with ESKD. Medicare costs per person per year range from $32,914 for KT patients, to $66,751 on peritoneal dialysis, to $87,561 for hemodialysis. This amount does not include the money paid by private health insurers as well as other sources of public health coverage such as the VA and state funds or Medicaid. Although about 90% of that cost goes toward dialysis treatment as the most popular modality for ESKD treatment, kidney transplantation (KT) is the optimal treatment for end-stage kidney disease (ESKD). It reduces mortality, improves quality of life, and is less costly than dialysis. Patients who can get a KT before starting dialysis, fare better post-transplant than those who are transplanted after they have started dialysis. Further, living donor KT (LDKT) is better than deceased donor KT (DDKT) because: (a) patients who can identify a living donor (LD) will get a KT much more quickly than ones awaiting DDKT7, and, (b) LDKT yields better outcomes than DDKT by improving cost effectiveness, reducing morbidity, and increasing long-term survival.

Research has shown significant disparities in ESKD for members of vulnerable groups (e.g., Hispanic/Latino, Native Americans, low income), and that African Americans (AA) are a particularly vulnerable group. The AA population is disproportionately represented among patients with ESKD. Although AAs represent only 13% of the US population, they represent over 30% of those with ESKD. Since the late 1970s the incidence of ESKD increased at a fourfold rate among AA compared with whites (WH). Kidney disease is particularly problematic because its major causes are diabetes and hypertension, two diseases that are more prevalent among AA and are related to a combination of physiological, lifestyle, behavioral, socioeconomic, and healthcare access differences between AA and WH. AA race is associated with: (a) lower likelihood of referral for KT among dialysis patients, (b) a longer time to complete evaluation for KT, (c) lower likelihood of getting a KT, (d) lower rates of pre-emptive listing for KT and, (e) lower rates of LDKT versus DDKT. Therefore, two of the best ways to reduce disparities in KT may be to increase (a) the number of vulnerable group members who complete KT evaluation and (b) the rate of LDKT. Our study is a two-pronged approach to address these two critical areas leading to disparities.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have scheduled a kidney transplant evaluation appointment at the Starzl Transplant Institute at the University of Pittsburgh Medical Center.
* Male or female
* English speaking
* ESKD patients aged 18 and over
* Patient has not previously received a kidney transplant
* Patient has not been accepted for kidney transplant in another center

Exclusion Criteria:

* Prior kidney transplant (excluded to eliminate the possibility that past experiences would affect their current treatment decisions)
* Patient is already on the United Network for Organ Sharing (UNOS) waiting list through another center
* Children under age 18 will be excluded because they have dissimilar underlying conditions, response patterns and decision-making authority as a result of their developmental stage and dependency on adult guardians.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1315 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Receipt of Kidney Transplant | Assessed via Post- transplant medical record review. An average time period to receive transplant and assess this outcome is approximately 43.6 months from baseline.
  This measure will assess whether or not the patient receives a kidney transplant

SECONDARY OUTCOMES:
Time to complete transplant evaluation | Assessed via medical record at completion of KT evaluation (Time 2) which can take up to one year from baseline
  We will use medical record data to measure the time from initiation of pre-KT workup to completing of kidney transplant evaluation
Kidney Transplant Decision Making (assessed using increasing levels of preference for a living versus deceased donor) | Assessed twice. First at initiation of pre-KT workup (Time 1) which is baseline. And next at the completion of evaluation (Time 2) which can take place up to one year from baseline.
  Kidney transplant decision making will be assessed using increasing levels of preference for a living versus deceased donor with 7 items adapted from the Kidney Transplant Questionnaire.
Booklet and video helpfulness (assess perceptions of the quality and helpfulness of the video and booklet) | Assessed at completion of evaluation (Time 2) which can take place up to one year from baseline.
  For participants in the TALK condition, we will assess perceptions of the quality and helpfulness of the video and booklet.
Quality of Life (KDQOL-SF) | Assessed at completion of evaluation (Time 2) which can take place up to one year from baseline.
  We will use the KDQOL-SF to measure QOL. The SF-36 serves as the generic core of this measure. The KDQOL also includes items relevant to patients with kidney disease.
Type of transplant (whether the patient receives a Living or Deceased Donor Kidney Transplant) | Assessed via Post- transplant medical record review. An average time period to receive transplant and assess this outcome is approximately 43.6 months from baseline.
  This measure will assess whether the patient receives a Living or Deceased Donor Kidney Transplant

CONTACTS AND LOCATIONS:
Overall Officials: Mary Amanda Dew, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Myaskovsky L, Leyva Y, Puttarajappa C, Kalaria A, Ng YH, Velez-Bermudez M, Zhu Y, Bryce C, Croswell E, Wesselman H, Kendall K, Chang CC, Boulware LE, Tevar A, Dew MA. Kidney Transplant Fast Track and Likelihood of Waitlisting and Transplant: A Nonrandomized Clinical Trial. JAMA Intern Med. 2025 May 1;185(5):499-509. doi: 10.1001/jamainternmed.2025.0043. PMID 40063052